CLINICAL TRIAL: NCT05682820
Title: Analysis of Radiological Features of Lateral Femoral Impaction Fracture / Lateral Femoral Notch Sign
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Head of the Clinic, Artromedical Konrad Malinowski Clinic
Other Study IDs: 1-rad-ar-2023
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ACL tear: Patients with ACL tear- MRIs will be assessed
  Interventions: Diagnostic Test: Measurements on knee MRI performed during routine clinical practice
- Patients without ACL tear: Patients without ACL tear - MRIs will be assessed
  Interventions: Diagnostic Test: Measurements on knee MRI performed during routine clinical practice

INTERVENTIONS:
Diagnostic Test: Measurements on knee MRI performed during routine clinical practice — Patients after knee injury are often advised to undergo knee MRI for diagnosis. Measurements on knee MRI performed during routine clinical practice will be made.

SUMMARY:
Analysis of Radiological Features of Lateral Femoral Impaction Fracture (LFC-IF) / Lateral Femoral Notch Sign will be performed on MRIs of consecutive patients after anterior cruciate ligament (ACL) injuries and without ACL injuries.

DETAILED DESCRIPTION:
Two independent measurers will twicely measure the radiological features of Lateral Femoral Impaction Fracture / Lateral Femoral Notch Sign on MRIs of consecutive patients after anterior cruciate ligament (ACL) injuries and without ACL injuries. In cases without ACL injuries, radiological features of terminal sulcus (TS), a native sulcus located on the lateral femoral condyle, will be measured. Intra- and inter-rater agreements will be calculated.

The following radiological features will be assessed/ measured:

1. Presence of LFC-IF/ TS
2. LFC-IF/ TS depth
3. LFC-IF/ TS length
4. Distance from Blumensaat line to the front border of LFC-IF / TS
5. Distance from Blumensaat line to the deepest part of LFC-IF / TS
6. Distance from Blumensaat line to the rear border of LFC-IF / TS

ELIGIBILITY:
Inclusion Criteria:

* Performed knee MRI with or without ACL tear

Exclusion Criteria:

* Osteophytes hindering assessment of LFC-IF/ TS morphology
* Morphological disturbances hindering assessment of LFC-IF/ TS morphology

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients with knee MRI with or without ACL tear, aged 18-45 years old, all sexes, with eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Distance from Blumensaat line to the rear border of LFC-IF / TS | At the time of MRI exam
  Distance from Blumensaat line to the rear border of LFC-IF /TS

SECONDARY OUTCOMES:
Distance from Blumensaat line to the deepest part of LFC-IF / TS | At the time of MRI exam
  Distance from Blumensaat line to the deepest part of LFC-IF / TS
Distance from Blumensaat line to the front border of LFC-IF / TS | At the time of MRI exam
  Distance from Blumensaat line to the front border of LFC-IF / TS
LFC-IF / TS length | At the time of MRI exam
  LFC-IF / TS length
LFC-IF / TS depth | At the time of MRI exam
  LFC-IF / TS depth
Presence of LFC-IF / TS | At the time of MRI exam
  Presence of LFC-IF / TS

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lodewijks PCAM, Delawi D, Bollen TL, Dijkhuis GR, Wolterbeek N, Zijl JAC. The lateral femoral notch sign: a reliable diagnostic measurement in acute anterior cruciate ligament injury. Knee Surg Sports Traumatol Arthrosc. 2019 Feb;27(2):659-664. doi: 10.1007/s00167-018-5214-x. Epub 2018 Oct 13. PMID 30317524
- [Result] Wierer G, Simetinger T, Hudelmaier M, Moroder P, Hoffelner T. Fate of the lateral femoral notch following early anterior cruciate ligament reconstruction. Knee. 2020 Mar;27(2):414-419. doi: 10.1016/j.knee.2020.01.009. Epub 2020 Feb 7. PMID 32037234
- [Result] Dimitriou D, Reimond M, Foesel A, Baumgaertner B, Zou D, Tsai TY, Helmy N. The deep lateral femoral notch sign: a reliable diagnostic tool in identifying a concomitant anterior cruciate and anterolateral ligament injury. Knee Surg Sports Traumatol Arthrosc. 2021 Jun;29(6):1968-1976. doi: 10.1007/s00167-020-06278-w. Epub 2020 Sep 24. PMID 32974801
- [Result] Bernholt DL, DePhillipo NN, Grantham WJ, Crawford MD, Aman ZS, Kennedy MI, LaPrade RF. Morphologic Variants of Posterolateral Tibial Plateau Impaction Fractures in the Setting of Primary Anterior Cruciate Ligament Tear. Am J Sports Med. 2020 Feb;48(2):318-325. doi: 10.1177/0363546519893709. Epub 2020 Jan 3. PMID 31899869
- [Result] Bernholt DL, DePhillipo NN, Crawford MD, Aman ZS, Grantham WJ, LaPrade RF. Incidence of Displaced Posterolateral Tibial Plateau and Lateral Femoral Condyle Impaction Fractures in the Setting of Primary Anterior Cruciate Ligament Tear. Am J Sports Med. 2020 Mar;48(3):545-553. doi: 10.1177/0363546519895239. Epub 2020 Jan 9. PMID 31917606